CLINICAL TRIAL: NCT00369291
Title: CPG 7909 Oligodeoxynucleotides (ODNS) After Autologous Transplantation to Enhance Immune Reconstitution
Brief Title: CpG 7909 in Treating Patients Who Have Undergone Autologous Stem Cell Transplant
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003LS014; UMN-0302M41542 (Other: IRB, University of Minnesota); UMN-MT2003-03 (Other: Blood and Marrow Transplantation Program)
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Germ Cell Tumor; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell | interventions — keyhole-limpet hemocyanin; Tetanus Toxoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CpG 7909 (Experimental): Patients treated with CpG 7909 oligodeoxynucleotides (ODNs) after autologous transplantation to enhance immune reconstitution.
  Interventions: Biological: keyhole limpet hemocyanin; Biological: tetanus toxoid

INTERVENTIONS:
Biological: keyhole limpet hemocyanin — KLH is a foreign protein to humans, it will be used to assess the immune response to a neo-antigen given as a single injection, 1 mg subcutaneously in the arm (per MT1999-06).
  Other Names: KLH
Biological: tetanus toxoid — Tetanus toxoid booster 0.5 ml intramuscularly (IM) in the opposite arm (per MT1999-06)

SUMMARY:
RATIONALE: Giving CpG 7909 after an autologous stem cell transplant may make a stronger immune response and prevent or delay the recurrence of cancer.

PURPOSE: This phase I trial is studying the side effects and best dose of CpG 7909 in treating patients who have undergone autologous stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether CpG 7909 enhances immune function, as measured by the response to keyhole limpet hemocyanin (neo-antigen) and tetanus toxoid (memory antigen), in patients who have undergone autologous stem cell transplantation.

Secondary

* Determine if dose escalation of CpG 7909, within a range of previously tested safe doses of CpG 7909, impacts upon the primary immune readouts.

OUTLINE: This is a non-randomized, dose-escalation study of CpG 7909.

Patients receive CpG 7909 subcutaneously (SC) on days 1, 7, and 14. Patients receive keyhole limpet hemocyanin SC and tetanus toxoid SC on day 7.

Cohorts of 3-6 patients receive escalating doses of Cp6 7909 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. A total of 10 patients are treated at the MTD.

Blood is collected at baseline and at approximately day 40 for immunological studies, including immunoenzyme techniques, antibody response assays, and immunophenotyping.

After completion of study treatment, patients are followed every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have undergone autologous transplantation for non-Hodgkin's lymphoma (NHL), Hodgkin's disease, acute myelogenous leukemia (AML), germ cell tumors, or multiple myeloma.
* Patients must be eligible for and consent to participate in study MT1999 06 - Vaccination with tetanus toxoid and Keyhole Limpet Hemocyanin (KLH) to assess antigen specific immune responses (BB-IND 10430).
* Patients will be eligible to receive CpG 7909 and vaccines on or after day 60 post transplant. No patients are eligible for this protocol beyond day 74 post transplant. Therefore, all patients will start therapy on this protocol between days 60-74 post transplant to allow for patient scheduling flexibility.
* Patients must have engraftment and be independent of transfusion support or growth factor support.
* Patients must not have received platelet or red-cell transfusions in the previous week.
* Patients must have been continuously off all growth factors for at least 1 week.
* Unsupported counts must be:

  * platelets ≥ 50,000/ml
  * Hgb ≥ 9 gm/ul
  * Absolute neutrophil count ≥ 1000/µL
  * Absolute lymphocyte count ≥ 500/µL
* Patients must have a current performance status of 0-1 (Eastern Cooperative Oncology Group) or 70-100% (Karnofsky.
* Patients must be afebrile, off antibiotics therapeutic (not prophylactic), and free of evidence of active infection. Patients must be off intravenous (IV) hyperalimentation and IV fluids.
* Minimum laboratory values within 2 weeks of entry: Creatinine ≤ 2.0 mg/dl or CrCl ≥ 50 ml/min, Bilirubin, ALT ≤ 2 x normal
* Age >18 years
* Patients receiving or scheduled to receive planned radiation therapy, growth factor therapy, or steroid therapy during the study period will be ineligible. Patients must have completed all planned post-transplant radiation therapy if applicable.
* Patients must be able to give written informed consent and agree to comply with the study parameters
* Patients must agree to use contraception during the study.

Exclusion Criteria:

Patients with one or more of the following:

* Active infection, or fever >38.2˚C
* Significant nonmalignant disease including documented HIV infection, uncontrolled hypertension (diastolic blood presses >115 mmHg), unstable angina, congestive heart failure (NY Class II), poorly controlled diabetes, coronary angioplasty within 6 months, myocardial infarction with the last 6 months, or uncontrolled atrial or ventricular cardiac arrhythmias.
* Hematopoietic growth factors administered within 1 week of study entry.
* Expected to require additional cytotoxic therapy within 30 days of study
* Receiving other post-transplant investigational agents
* Patients with a history of autoimmune diseases will be ineligible for this protocol
* It is unknown whether CpG 7909 may exacerbate autoimmune disorders by its immunomodulatory effects. Therefore, subjects with a history of autoimmune disease should not receive CpG 7909. Controlled thyroid disease is permissible.
* Systemic corticosteroids or other immunosuppressants
* Pregnant or lactating (It is unlikely and probably unwise that a women of childbearing potential become pregnant this early after transplant, however; if any suspicion, a pregnancy test should be done)
* Not meeting one or more of the eligibility criteria, as listed above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2003-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Enhanced immune function as measured by response to keyhole limpet hemocyanin and tetanus toxoid | 1 Month after vaccine
  anti-KLH IgG

SECONDARY OUTCOMES:
Impact of dose escalation of CpG 7909 on primary immune readouts | At study completion
  Compare primary outcome between cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Marcie Tomblyn, MD, MS, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States